CLINICAL TRIAL: NCT06446739
Title: LoW Dose-Intensity vs. Standard Dose-Intensity COntinuous Renal ReplaceMent Therapy in Critically Ill Patients (WISDOM): A Pilot Randomized Trial
Brief Title: LoW Dose-Intensity vs. Standard Dose-Intensity COntinuous Renal ReplaceMent Therapy in Critically Ill Patients (WISDOM)
Acronym: WISDOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00140224
Record Dates: First submitted 2024-04-16; First posted 2024-06-06 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury; Dialysis; Complications
Keywords: acute kidney injury; continuous renal replacement therapy; dose-intensity; randomized trial; pilot feasibility
MeSH Terms: conditions — Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Low dose-intensity (Experimental): The intervention arm will consist of low dose-intensity CRRT, defined as the hourly delivery of a total effluent of 10-15 mL/kg/hr while receiving CRRT. The intervention dose-intensity is based on the rationale that 10-15 mL/kg/hr is the lower threshold of dose-intensity currently provided in clinical practice and prior observational data showing this threshold is tolerated and safe.
  Interventions: Device: Continuous Renal Replacement Therapy (CRRT)
- Standard dose-intensity (Active Comparator): The control arm will receive a dose-intensity CRRT of 25-30 mL/kg/hr while receiving CRRT, aligned with local practice and information by international clinical practice guidelines. The control dose-intensity is based on the rationale that this is currently recommended in clinical practice guidelines and is commonly applied in routine practice.
  Interventions: Device: Continuous Renal Replacement Therapy (CRRT)

INTERVENTIONS:
Device: Continuous Renal Replacement Therapy (CRRT) — Continuous Renal Replacement Therapy (CRRT) is a continuous form of acute renal replacement (hemofiltration/dialysis) therapy provided to critically ill patients with multi-organ dysfunction receiving life support in the intensive care unit (ICU).

SUMMARY:
An estimated 10-15% of critically ill patients with acute kidney failure in the intensive care unit receive acute dialysis therapy. The majority of these patients initially receive a continuous form of dialysis therapy call continuous renal replacement therapy (CRRT). Prior studies have suggested that higher CRRT dose-intensity improved health outcomes for these patients; however, this was not found in high-quality clinical trials. These more recent trials suggested a lower range of dose-intensity compared with the higher range as the new standard of care. This was incorporated into guidelines. To date, no clinical trials have evaluated this lower range and specifically, it is plausible that an even lower dose-intensity of CRRT may be well tolerated, safe, associated with similar outcomes and be more cost-effective. This is the objective of the WISDOM trial, to compare the guideline standard with lower dose-intensity among patients who are started on CRRT in the intensive care unit.

DETAILED DESCRIPTION:
Purpose: To primarily determine whether a lower CRRT dose-intensity in critically ill patients with acute kidney injury (AKI) is non-inferior to standard CRRT dose-intensity and to secondarily determined whether lower CRRT dose intensity will shorten total CRRT duration and improve kidney recovery compared with standard CRRT dose-intensity.

Hypothesis: The primary hypothesis of the WISDOM trial is that lower CRRT dose-intensity is non-inferior to current standard guideline-directed CRRT dose-intensity for critically ill patients with AKI with respect to duration of CRRT and successful liberation from RRT and kidney recovery. The secondary hypothesis of the WISDOM trial is that lower dose-intensity is superior to current standard guideline-directed CRRT dose-intensity for critically ill patients with AKI with respect to duration of CRRT and successful liberation from RRT and kidney recovery.

Justification: No randomized controlled trial (RCT) to date has specifically evaluated the lower dose-intensity threshold for critically ill patients receiving CRRT. Specifically, there has been no specific evidence or guidance on the minimum dose-intensity targets for patients receiving CRRT. This is important for several reasons. First, CRRT is an invasive, resource intensive and expensive therapy. As such, there should be a concerted effort to minimize time on RRT and facilitate early recovery and weaning. Second, abundant evidence derived from secondary analyses have suggested that higher CRRT dose-intensity can propagate oliguria, prolong CRRT therapy and delay kidney recovery. This would imply that lower dose-intensity may facilitate kidney recovery and earlier weaning from CRRT. Third, there may be added implications of higher dose-intensity, including prolongation of non-renal organ support, such as delay in weaning from invasive mechanical ventilation. Fourth, evidence derived from observational registries show that lower CRRT dose-intensity, in the range proposed in this trial, provides comparable efficacy in azotemic, metabolic and acid-base homeostasis with similar outcomes. Observational data have suggested a prescribed CRRT dose-intensity of 15 mL/kg/hr may be sufficient for metabolic and azotemic control and is not associated with worse outcomes compared with guideline directed dose-intensity. This is lower quality evidence, however, implies that lower dose-intensity may be acceptable and safe. Fifth, it is plausible that following a short period of metabolic stabilization with CRRT, the minimum recommended CRRT dose-intensity of 20-25 mL/kg/hr may be excessive and have unmeasurable harm (e.g., excessive clearance of electrolytes, micronutrients, and medications [antimicrobials]). Finally, the prescription of a lower CRRT dose-intensity may have meaningful impact on reducing bedside nursing workload (e.g., fewer replacement solution bag changes) and reducing costs attributable to CRRT (e.g., lower effluent rates will reduce total replacement solution utilized).

While this proposal outlines a pilot feasibility trial, it is aimed at performing a larger rigorous RCT that will generate generalizable and high-quality evidence to impact clinical practice. The findings of the main phase of the WISDOM trial will provide clearer evidence to guide the prescription of a minimal dose-intensity for patients receiving CRRT. While this may be an effluent dose of 20-25 mL/kg/hr, it is entirely plausible that this will be a lower dose-intensity.

Objectives: The overall WISDOM trial program will address whether a lower CRRT dose-intensity in critically ill patients with AKI is non-inferior to standard CRRT dose-intensity and will secondarily address whether lower CRRT dose intensity will shorten total CRRT duration and improve kidney recovery compared with standard CRRT dose-intensity.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* weight ≥ 55 kg
* plan to initiate CRRT or within 24 hours of having started CRRT for AKI
* expected to survive and receive CRRT for a duration of ≥ 48 hours
* able to provide informed consent or have an authorized representative provide consent after being informed on the details and risks of the trial unless a deferred consent process is approved by local Research Ethics Board (REB).

Exclusion Criteria:

* indication for sustained higher dose-intensity CRRT as designated by the attending clinicians
* end-stage kidney disease receiving maintenance dialysis
* receipt of any RRT for AKI during the current hospitalization
* inability to comply with the requirements of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Difference in delivered CRRT dose-intensity | Through study completion, an average of 1 month.
  This pilot trial will target detection of a minimum difference of 10 mL/kg/hr in delivered dose-intensity.

SECONDARY OUTCOMES:
Feasibility - consent rate | Through study completion, at 90-days.
  Consent rate for participation by patient or surrogate decision-maker (SDM).
Feasibility - time to enrollment | During active recruitment into the trial, approximately 1 year.
  Time from eligibility (e.g., starting RRT) to randomization.
Feasibility - adherence to prescribed CRRT dose-intensity | Through study completion, at 90-days.
  Protocol adherence for allocated CRRT dose-intensity.
Feasibility - ascertainment to delivered CRRT process measures | Through study completion, at 90-days.
  Ability to capture delivered CRRT dose-intensity measures.
Feasibility - outcome ascertainment | Through study completion, at 90-days.
  Ability to capture patient and kidney endpoints at 90-days.
Feasibility - recruitment rate | During active recruitment into the trial, approximately 1 year.
  Ability to recruit 2 patients per site per month.

OTHER OUTCOMES:
Daily bicarbonate while receiving CRRT, an average of 1 month. | Through study completion, at 90-days.
  Physiological and biochemical outcomes.
Daily serum phosphate while receiving CRRT, an average of 1 month | Through study completion, at 90-days.
  Physiological and biochemical outcomes.
Daily serum urea while receiving CRRT, an average of 1 month | Through study completion, at 90-days.
  Physiological and biochemical outcomes.
The total treatment time per day while receiving CRRT following randomization. | Through study completion, at 90-days.
  Process of care measures.
The total number of hemofilter/circuit replacements while receiving CRRT following randomization. | Through study completion, at 90-days.
  Process of care measures.
The lowest and highest CRRT dose-intensity delivered for any given hour following randomization. | While receiving CRRT, an average of 1 month.
  Process of care measures.
The proportion of hours of CRRT when the dose-intensity is in the target range following randomization. | Through study completion, at 90-days.
  Process of care measures.
Occurrence of adverse and serious adverse events. | Through study completion, at 90-days.
  Safety measures.
Occurrence of adverse events and serious adverse events leading to discontinuation of the trial intervention. | Through study completion, at 90-days.
  Safety measures.
RRT-free days at 90-days. | Through study completion, at 90-days.
  Clinical Outcomes.
The total volume of replacement/dialysate fluid used per day following randomization. | Through study completion, at 90-days.
  Process of care measures
The total number of doses of supplemental electrolytes administered while receiving CRRT following randomization. | Through study completion, at 90 days.
  Process of care measures
The cumulative doses of supplemental electrolytes administered while receiving CRRT following randomization. | Through study completion, at 90 days.
  Process of care measures
The mean daily net ultrafiltration delivery while receiving CRRT following randomization. | Through study completion, at 90 days.
  Process of care measures

CONTACTS AND LOCATIONS:
Overall Officials: Sean M Bagshaw, MD, Principal Investigator — University of Alberta; Ron Wald, Principal Investigator — St. Michael's Hospital (Unity Health)
Locations (4):
- Canada (4):
  - University of Alberta Hospital, Edmonton, Alberta
  - Hamilton General Hospital, Hamilton, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Regina General Hospital/Saskatchewan Health Authority, Regina, Saskatchewan

REFERENCES:
- [Derived] Beaubien-Souligny W, Thompson Bastin M, Teixeira JP, Cerda J, Connor MJ Jr, Dijanic Zeidman A, Garimella PS, Juncos L, Lopez-Ruiz A, Mehta R, Reis T, Rizo-Topete L, Silver SA, Da Silva JR, Speer R, Vijayan A, Wells C, Wille K, Yessayan L, Tolwani A, Neyra JA. Proceedings of the University of Alabama at Birmingham Continuous Renal Replacement Therapy Academy (2023-2024): Managing De-Escalation of Acute Renal Replacement Therapy and Optimizing Drug Dosing during Renal Replacement Therapy Transitions. Kidney360. 2025 Oct 1;6(10):1798-1809. doi: 10.34067/KID.0000000951. Epub 2025 Aug 8. PMID 40779331